CLINICAL TRIAL: NCT00738101
Title: Compassionate Use of an Intravenous Fat Emulsion Comprised of Fish Oil in the Treatment of Parenteral Nutrition Induced Liver Injury in Infants
Brief Title: Compassionate Use of an Intravenous Fish Oil Emulsion in the Treatment of Liver Injury in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Muralidhar Premkumar, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23365
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Cholestasis; Cholestasis of Parenteral Nutrition
Keywords: Omega-3; Omegaven; Cholestasis; Liver damage
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides

STUDY DESIGN:
Intervention Model Description: Initiation of Study is defined as the day the Fish Oil Emulsion was initiated.
  End of Study (EOS) is defined as discontinuation of fish oil emulsion, death, transplant, or discharge from the hospital.
  In infants who meet the eligibility criteria for Fish Oil Emulsion arm will receive Fish Oil Emulsion after enrollment under the study. Therapy with Fish Oil Emulsion (Omegaven) will be provided at a dose of 1 gm/kg/day (by continuous infusion) and will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. If previously on Intralipid, it will be stopped prior to initiation of Fish Oil Emulsion.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fish Oil Emulsion Arm (Experimental): In infants who meet the eligibility criteria for Fish Oil Emulsion arm will receive Fish Oil Emulsion after enrollment under the study.
  Therapy with Fish Oil Emulsion (Omegaven) will be provided at a dose of 1 gm/kg/day (by continuous infusion) and will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. If previously on Intralipid, it will be stopped prior to initiation of Fish Oil Emulsion.Fish oil emulsion will be provided as a continuous intravenous emulsion over 24 hours.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Therapy with Omegaven will be provided at a dose of 1 gm/kg/day (by continuous infusion). Omegaven will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. Treatment will be given for as long as the child needs any TPN AND has a conjugated bilirubin greater than 2 mg/dL for a maximum of 5 years. If the infant no longer is requiring any TPN, then the Omegaven will be stopped regardless of bilirubin. If the bilirubin is less than 2 mg/dL but the child still requires TPN, then the Omegaven will be continued until the infant no longer requires TPN.
  Other Names: Omega-3 enriched fat emulsion

SUMMARY:
To provide a mechanism for critically ill infants with parenteral nutrition (PN) associated cholestasis to receive Omegaven for compassionate use situations for which there are no satisfactory alternative treatments.

DETAILED DESCRIPTION:
Inpatient Use of Omegaven:

Each family will have the severity of their child's condition explained to them and the available data regarding the benefit of the novel preparation explained using the preliminary safety and efficacy data from Boston Children's Hospital and TCH. Families will have the potential risks and benefits of the product explained. The lack of long-term follow-up information regarding the effects of Omegaven will be discussed.

Bottles containing 50mL or 100 mL of 10% Omegaven will be purchased from International Pharmacy of Hamburg, Germany. Omegaven is manufactured by Fresenius Kabi AG, Bad Homburg v.d.h, Germany. Omegaven is formulated as an emulsion from fish oils. The family (or legal guardian) will be billed for the Omegaven as part of their hospital bill from Texas Children's Hospital.

Omegaven will be dispensed per Texas Children's Hospital policy and procedures for fat emulsions.

All study materials will be stored securely until the time of administration. The bottles will be stored at room temperature below 30° C (do not freeze). Damaged or suspect drug will be returned unused to Fresenius- Kabi. Containers should be shaken before use.

All supplies for the study will be accompanied by accountability and shipping documents and will be maintained by the Investigator or deputy (e.g. research pharmacist). Information recorded on these accountability and shipping documents will include relevant dates, batch numbers, quantities received or dispensed, to whom dispensed, returned drug, and drug lost or damaged. At the end of the study, all used and unused Omegaven will be accounted for. If expired, the remaining drug supplies will be destroyed.

Details of Omegaven Administration:

Therapy with Omegaven will be provided at a dose of 1 gm/kg/day (by continuous infusion). Omegaven will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. Parenteral fat emulsion (Intralipid) will be administered only if necessary to administer adequate calories during Omegaven therapy. The same standards of care provided to all patients receiving parenteral nutrition solution will be followed.

Ongoing monitoring during therapy related to safety and efficacy:

Safety will be assessed using the following outcome variables.

First, we will calculate the number (total and daily rate) of bloodstream infections prior to therapy. We will monitor this rate in each baby receiving Omegaven and compare with the previous rate. Currently, the rate of infection in infants receiving Omegaven is about half of the historical control rate at TCH.

Second, we will monitor growth rate using weight, length and head circumference growth. Growth will be compared both to the pre-treatment period and the expected rate of growth. We have established and have guidelines for optimal growth targets and management will be targeted on achieving these rates. We will monitor these carefully. For babies in the NICU or Level 2 nurseries, Dr. Abrams will supervise the nutritional management directly. Infants in the PICU or PCU will be followed by Dr. Carter with the critical care staff. This approach has been in place for the current group of 16 infants and growth has been excellent although final calculations are pending.

Third, we will monitor infants who are not receiving any enteral feeding at all for more than 4 weeks for any evidence of essential fatty acid (EFA) deficiency. Measurements will be repeated at the end of every 4 weeks that the subject remains without any enteral nutrition intake. Although the exact value suggestive of a deficiency is controversial, usually a level greater than 0.4 is considered evidence of EFA deficiency. This measurement may be made using 0.2 mL of serum in the lab of Dr. William Heird. Samples will be drawn monthly for infants who are NPO and run as a batch in Dr. Heird's lab in the CNRC every 6 months. Because data are not available for clinical use, we will include in the consent the possibility of EFA deficiency. We note again that no infant ever treated with Omegaven has ever shown clinical evidence of EFA deficiency, that very transient mild deficiency may occur in about 5% of infants and that there is no clinical intervention we would use in this case or that has ever been given without clinically apparent EFA deficiency.

Fourth, we will record and monitor the following lab and clinical results for the DSMB: electrolytes, calcium, phosphorus, magnesium, alkaline phosphatase, glucose, triglycerides, BUN, creatinine, conjugated and unconjugated bilirubin, albumin, prealbumin, CRP, WBC, RBC, platelets, PT, PTT, any evidence of bleeding, and positive blood cultures. These labs will be drawn as clinically relevant, not as a specific result of the study.

Finally, with regard to developmental follow-up we will indicate to families that all infants with cholestasis may be at risk for developmental delays and recommend that they be followed. There is no mechanism in place to assure this follow-up occurs for any infants in the TCH nurseries however.

Dose Modification

Hypertriglyceridemia:

If hypertriglyceridemia develops, defined as serum triglyceride levels > 300 mg/dL, the following will be considered prior to reducing the dose:

1. If the level was obtained while the patient was receiving a continuous 24- hour infusion of Omegaven, the total dose should be infused over 20 hours, and a repeat serum triglyceride level obtained prior to resuming the infusion 4 hours later.
2. Other sources of hypertriglyceridemia should be considered and addressed (drugs, renal disease)

If necessary if the triglycerides continue to remain high despite the aforementioned interventions, a dosage reduction of 25% will be considered.

Duration of Therapy

Patients will remain on Omegaven until weaned from PN.

In the event that a patient who has been listed for a liver or liver/intestinal transplant has an organ become available, the participation in this protocol will not preclude them from receiving the transplant. Omegaven will not be administered post transplant.

Treatment will be given for as long as the child needs any TPN AND has a conjugated bilirubin greater than 2 mg/dL for a maximum of 5 years. If the infant no longer is requiring any TPN, then the Omegaven will be stopped regardless of bilirubin. If the bilirubin is less than 2 mg/dL but the child still requires TPN, then the Omegaven will be continued up to a total of 5 years or whenever the infant no longer requires TPN. The reason for stopping Omegaven when the infant no longer requires TPN is that this would be the only reason many infants would still need IV access and therefore the risk of maintaining IV access only for the medication is likely to exceed the benefit of Omegaven at that point.

Legal and Ethics Requirements:

This study has been approved by the BCM IRB under a FDA Investigational New Drug Application using IND #102,843.

The Investigators will be responsible for obtaining an Informed Consent signed by each patient or his/her legally authorized representative prior to his/her participation in the study in accordance with the Code of Federal Regulations, Title 21, Part 50.20. Informed Consent will be obtained from a patient or his/her legally authorized representative after a full explanation of the purpose of the study, the risks and discomforts involved, potential benefits, etc. have been provided by the Investigator or designee, both verbally and in writing. The person who signed the consent will be given a copy of the signed consent form. The lack of long-term follow-up information regarding the effects of Omegaven will be discussed.

Home Use of Omegaven:

In order for a subject to receive the Omegaven® at home through the home health care agency, subjects will first be required to be admitted to Texas Children's Hospital for 72 hours in initiate the administration of the Omegaven®. This will allow time for observation of any unexpected side effects and for parents to be provided education on home TPN and Omegaven®.

If a subject has already received Omegaven® either at TCH or at another hospital, they will not be required to be admitted for the 72 hour inpatient admission prior to starting Omegaven® at home. Parent training will occur during the previous hospital admission and will continue through the TCH Pediatric Intestinal Rehabilitation Clinic.

This population will include infants up to 5 years of age. The Omegaven® dose for home use will be the same as that used while in the hospital: 1 gm/kg/day. As with the inpatient part of the protocol, this is a maximum dose and may be decreased at the discretion of the TCH Pediatric Intestinal Rehabilitation Clinic Team.

Outpatient Monitoring:

After the initial evaluation by the TCH Pediatric Intestinal Rehabilitation Clinic physicians, subjects will return to the clinic for routine follow-up. Subjects will be asked to return to the clinic every 2 weeks for the first 2 months of treatment. Thereafter, subjects will return to the clinic on a monthly basis, or as directed by the clinic team. Orders for home use of Omegaven® will be signed by the physician at the clinic visits, ensuring that subjects are compliant with study parameters while receiving the treatment drug.

Routine monitoring done at clinic appointments and at home will be recorded for study purposes and data collection. No blood work will be done for study purposes only. Lab monitoring will typically be done every week to two weeks at home and at each clinic visit.

FDA Contact:

Division of Gastroenterology and Inborn Errors Products Division of Drug Information (DDI) (855) 543-3784 or (301) 796-3400; druginfo@fda.hhs.gov

ELIGIBILITY:
Inclusion Criteria:

* Be greater than 14 days old and less than 5 years old
* Conjugated bilirubin greater than 2 mg/dL.
* Be expected to require intravenous nutrition for at least an additional 28 days

Exclusion Criteria:

* Have a congenitally lethal condition (e.g. Trisomy 13).
* Have clinically severe bleeding not able to be managed with routine measures.
* Have evidence of a viral hepatitis or primary liver disease as the primary etiology of their cholestasis.
* Have other health problems such that survival is extremely unlikely even if the infant's cholestasis improves.

Home Use of Omegaven®:

In order for a subject to receive the Omegaven® at home through a home health care agency, subjects will first be required to be admitted to Texas Children's Hospital for 72 hours in initiate the administration of the Omegaven®. This will allow time for observation of any unexpected side effects and for parents to be provided education on home TPN and Omegaven®.

If a subject has already received Omegaven® either at TCH or at another hospital, they will not be required to be admitted for the 72 hour inpatient admission prior to starting Omegaven® at home. Parent training will occur during the previous hospital admission and will continue through the TCH Pediatric Intestinal Rehabilitation Clinic.

Outpatient Monitoring:

After the initial evaluation by the TCH Pediatric Intestinal Rehabilitation Clinic physicians, subjects will return to the clinic for routine follow-up. Subjects will be asked to return to the clinic every 2 weeks for the first 2 months of treatment. Thereafter, subjects will return to the clinic on a monthly basis, or as directed by the clinic team.

Ages: 14 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2008-09; Primary Completion 2019-03-27 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murali Premkumar, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Please see the IPD sharing section below.

REFERENCES:
- [Background] Dudrick SJ, Wilmore DW, Vars HM, Rhoads JE. Long-term total parenteral nutrition with growth, development, and positive nitrogen balance. Surgery. 1968 Jul;64(1):134-42. No abstract available. PMID 4968812
- [Background] Wilmore DW, Dudrick SJ. Growth and development of an infant receiving all nutrients exclusively by vein. JAMA. 1968 Mar 4;203(10):860-4. No abstract available. PMID 4965871
- [Background] Mullick FG, Moran CA, Ishak KG. Total parenteral nutrition: a histopathologic analysis of the liver changes in 20 children. Mod Pathol. 1994 Feb;7(2):190-4. PMID 8008742
- [Background] Freund HR. Abnormalities of liver function and hepatic damage associated with total parenteral nutrition. Nutrition. 1991 Jan-Feb;7(1):1-5; discussion 5-6. PMID 1802177
- [Background] Beath SV, Davies P, Papadopoulou A, Khan AR, Buick RG, Corkery JJ, Gornall P, Booth IW. Parenteral nutrition-related cholestasis in postsurgical neonates: multivariate analysis of risk factors. J Pediatr Surg. 1996 Apr;31(4):604-6. doi: 10.1016/s0022-3468(96)90507-2. PMID 8801324
- [Background] Greenberg GR, Wolman SL, Christofides ND, Bloom SR, Jeejeebhoy KN. Effect of total parenteral nutrition on gut hormone release in humans. Gastroenterology. 1981 May;80(5 pt 1):988-93. No abstract available. PMID 6781979
- [Background] Yeh SL, Chen WJ, Huang PC. Effects of L-glutamine on induced hepatosteatosis in rats receiving total parenteral nutrition. J Formos Med Assoc. 1995 Oct;94(10):593-9. PMID 8527958
- [Background] Kubota A, Yonekura T, Hoki M, Oyanagi H, Kawahara H, Yagi M, Imura K, Iiboshi Y, Wasa K, Kamata S, Okada A. Total parenteral nutrition-associated intrahepatic cholestasis in infants: 25 years' experience. J Pediatr Surg. 2000 Jul;35(7):1049-51. doi: 10.1053/jpsu.2000.7769. PMID 10917294
- [Background] Moss RL, Das JB, Ansari G, Raffensperger JG. Hepatobiliary dysfunction during total parenteral nutrition is caused by infusate, not the route of administration. J Pediatr Surg. 1993 Mar;28(3):391-6; discussion 396-7. doi: 10.1016/0022-3468(93)90238-g. PMID 8468653
- [Background] Helms RA, Christensen ML, Mauer EC, Storm MC. Comparison of a pediatric versus standard amino acid formulation in preterm neonates requiring parenteral nutrition. J Pediatr. 1987 Mar;110(3):466-70. doi: 10.1016/s0022-3476(87)80519-x. No abstract available. PMID 3102712
- [Background] Moss RL, Haynes AL, Pastuszyn A, Glew RH. Methionine infusion reproduces liver injury of parenteral nutrition cholestasis. Pediatr Res. 1999 May;45(5 Pt 1):664-8. doi: 10.1203/00006450-199905010-00009. PMID 10231861
- [Background] Meehan JJ, Georgeson KE. Prevention of liver failure in parenteral nutrition-dependent children with short bowel syndrome. J Pediatr Surg. 1997 Mar;32(3):473-5. doi: 10.1016/s0022-3468(97)90609-6. PMID 9094021
- [Background] Whalen GF, Shamberger RC, Perez-Atayde A, Folkman J. A proposed cause for the hepatic dysfunction associated with parenteral nutrition. J Pediatr Surg. 1990 Jun;25(6):622-6. doi: 10.1016/0022-3468(90)90348-d. PMID 2113578
- [Background] Zamir O, Nussbaum MS, Bhadra S, Subbiah MT, Rafferty JF, Fischer JE. Effect of enteral feeding on hepatic steatosis induced by total parenteral nutrition. JPEN J Parenter Enteral Nutr. 1994 Jan-Feb;18(1):20-5. doi: 10.1177/014860719401800120. PMID 8164298
- [Background] Kaminski DL, Adams A, Jellinek M. The effect of hyperalimentation on hepatic lipid content and lipogenic enzyme activity in rats and man. Surgery. 1980 Jul;88(1):93-100. No abstract available. PMID 6104363
- [Background] Hultin M, Carneheim C, Rosenqvist K, Olivecrona T. Intravenous lipid emulsions: removal mechanisms as compared to chylomicrons. J Lipid Res. 1995 Oct;36(10):2174-84. PMID 8576643
- [Background] Qi K, Al-Haideri M, Seo T, Carpentier YA, Deckelbaum RJ. Effects of particle size on blood clearance and tissue uptake of lipid emulsions with different triglyceride compositions. JPEN J Parenter Enteral Nutr. 2003 Jan-Feb;27(1):58-64. doi: 10.1177/014860710302700158. PMID 12549600
- [Background] Nestel PJ. Effects of N-3 fatty acids on lipid metabolism. Annu Rev Nutr. 1990;10:149-67. doi: 10.1146/annurev.nu.10.070190.001053. No abstract available. PMID 2200461
- [Background] Chen WJ, Yeh SL, Huang PC. Effects of fat emulsions with different fatty acid composition on plasma and hepatic lipids in rats receiving total parenteral nutrition. Clin Nutr. 1996 Feb;15(1):24-8. doi: 10.1016/s0261-5614(96)80257-3. PMID 16843991
- [Background] Yeh SL, Chen WJ, Huang PC. Effects of fish oil and safflower oil emulsions on diet-induced hepatic steatosis in rats receiving total parenteral nutrition. Clin Nutr. 1996 Apr;15(2):80-3. doi: 10.1016/s0261-5614(96)80024-0. PMID 16844003
- [Background] Kinsella JE, Lokesh B, Broughton S, Whelan J. Dietary polyunsaturated fatty acids and eicosanoids: potential effects on the modulation of inflammatory and immune cells: an overview. Nutrition. 1990 Jan-Feb;6(1):24-44; discussion 59-62. No abstract available. PMID 2135755
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Strijbosch RA, Lee S, Arsenault DA, Andersson C, Gura KM, Bistrian BR, Puder M. Fish oil prevents essential fatty acid deficiency and enhances growth: clinical and biochemical implications. Metabolism. 2008 May;57(5):698-707. doi: 10.1016/j.metabol.2008.01.008. PMID 18442636
- [Derived] Gura KM, Calkins KL, Premkumar MH, Puder M. Use of Intravenous Soybean and Fish Oil Emulsions in Pediatric Intestinal Failure-Associated Liver Disease: A Multicenter Integrated Analysis Report on Extrahepatic Adverse Events. J Pediatr. 2022 Feb;241:173-180.e1. doi: 10.1016/j.jpeds.2021.10.030. Epub 2021 Oct 23. PMID 34695449
- [Derived] Gura KM, Premkumar MH, Calkins KL, Puder M. Fish Oil Emulsion Reduces Liver Injury and Liver Transplantation in Children with Intestinal Failure-Associated Liver Disease: A Multicenter Integrated Study. J Pediatr. 2021 Mar;230:46-54.e2. doi: 10.1016/j.jpeds.2020.09.068. Epub 2020 Oct 8. PMID 33038344
- [Derived] Gura K, Premkumar MH, Calkins KL, Puder M. Intravenous Fish Oil Monotherapy as a Source of Calories and Fatty Acids Promotes Age-Appropriate Growth in Pediatric Patients with Intestinal Failure-Associated Liver Disease. J Pediatr. 2020 Apr;219:98-105.e4. doi: 10.1016/j.jpeds.2019.12.065. Epub 2020 Feb 12. PMID 32059815
- [Derived] Premkumar MH, Carter BA, Hawthorne KM, King K, Abrams SA. High rates of resolution of cholestasis in parenteral nutrition-associated liver disease with fish oil-based lipid emulsion monotherapy. J Pediatr. 2013 Apr;162(4):793-798.e1. doi: 10.1016/j.jpeds.2012.10.019. Epub 2012 Nov 16. PMID 23164314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment to this compassionate use protocol began in September 2007. Patients were enrolled from mainly the inpatient and some from outpatient population at Texas Children's Hospital, Houston, Texas.
Pre-assignment Details: There was no wash-out or run-in period.
Groups:
- Fish Oil Emulsion Arm: In infants who meet the eligibility criteria for Fish Oil Emulsion arm received Fish Oil Emulsion (Omegaven) after enrollment under the study.
  Therapy with Fish Oil Emulsion (Omegaven) was provided at a dose of 1 gm/kg/day (by continuous infusion) and was infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. If previously on Intralipid, it was stopped prior to initiation of Fish Oil Emulsion.Fish oil emulsion. Treatment was given for as long as the child needed any TPN. If the infant no longer required any TPN, then the Omegaven was stopped. Omegaven was continued even after resolution of cholestasis, as long as the need for parenteral nutrition persisted.
Period: Overall Study
Arm/Group | Fish Oil Emulsion Arm
Started | 293
Completed | 286 (7 exclusions. 5 primary liver or unrelated disease, 1 died before Omegaven, 1 repeat enrollment)
Not Completed | 7
Not completed — Physician Decision | 5
Not completed — Death | 1
Not completed — Repeat enrollment | 1

BASELINE CHARACTERISTICS:
Population: Infants were included based on the eligible criteria as described.
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 286
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 286
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] — Age (in days) of the subjects at the time of initiation of Omegaven
  Days | 78.13 (129.6)
Age, Customized [Mean (Standard Deviation); unit: weeks] — Population: In the missing numbers, the gestational age at birth was not known.
  weeks
    Postmenstrual Age at time of initiation: number analyzed (Participants) | 265
    Postmenstrual Age at time of initiation | 40.3 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 110
  Not Hispanic or Latino | 161
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 62
  White | 186
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Number; unit: participants]
  United States | 286
Infants with Cholestasis [Count of Participants; unit: Participants] — Cholestasis is defined as serum conjugated bilirubin ≥ 2 mg/dL at the time of initiation of Fish Oil Emulsion (Omegaven).
  Participants | 286
Need for Parenteral Nutrition [Count of Participants; unit: Participants] — Infants who required parenteral nutrition either complete or partial at the time of initiation of Fish Oil Emulsion (Omegaven) due to feeding difficulties.
  Participants | 286
Gestational Age at Birth [Mean (Standard Deviation); unit: weeks] — Gestational Age at birth in weeks. Population: Gestational age at birth was not available in 19 infants.
  weeks
    number analyzed (Participants) | 267
    (all) | 29.71 (5)
Birth weight [Mean (Standard Deviation); unit: grams] — Birth weight (grams) Population: Birth weight was not available in 61 infants
  grams
    number analyzed (Participants) | 225
    (all) | 1429.7 (905.4)

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Parenteral Nutrition Associated Cholestasis Prior to End of Study
Description: Time in days from the initiation of fish oil emulsions (initiation of study) until resolution of cholestasis as defined by serum conjugated bilirubin≤ 2 mg/dL prior to EOS (end of study).
Time Frame: From initiation to end of study (End of Study : Discontinuation of Fish Oil Emulsion, Death, Transplant, or Discharge from the hospital, whichever is achieved first, up to 5 years).
Population: 210 out of 286 infants in the study demonstrated resolution of cholestasis prior to the end of study.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Fish Oil Emulsion Arm: Once eligible, Soybean Oil Emulsion was discontinued and Fish Oil Emulsion was commenced at 1 g/kg/d. Fish Oil Emulsion was provided as an infusion over 18-24 hours a day. Fish Oil Emulsion was provided in a dedicated peripheral or central venous access.
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 210
Days | 38.02 (23.9)

2. Primary Outcome: All Cause Mortality During the Study.
Description: To describe proportion of infants who died secondary to any cause, related or unrelated to Fish Oil Emulsion.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 286
Participants | 30

3. Primary Outcome: Growth Z-scores for Weight
Description: The Z-score indicated the number of standard deviations away from the mean. A weight Z-score of 0 is equal to the mean. A weight Z-score of ≤ -2 indicates an underweight status, while a weight Z-score of ≥ 2 indicates overweight or obese status.
Time Frame: as for outcome 1
Population: Out of 286 infants enrolled in the study, weight at the end of study was available only in 260 infants. Missing data: 26 infants.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 260
z-score | -1.48 (1.45)

4. Secondary Outcome: Number of Infants Who Achieve Resolution of Parenteral Nutrition Associated Cholestasis
Description: To describe the number of infants who achieved resolution of cholestasis following initiation of fish oil emulsion.
Time Frame: as for outcome 1
Population: Only 285 out of 286 infants were included in this analysis. One infant had conjugated bilirubin <2 mg/dL at the initiation of fish oil emulsion. This infant had been initiated on fish oil emulsion at another institute. Fish oil emulsion in this infant was provided as a continuation of care from another hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 285
Participants
  Resolution of Cholestasis | 210
  Unresolved Cholestasis | 75

5. Secondary Outcome: Number of Subjects With Platelet Count <100,000/µL
Description: To describe the number of study subjects who experienced a platelet count below <100,000/µL anytime during the duration of the study.
Time Frame: as for outcome 1
Population: Out of 286 infants enrolled in the study, weight at the end of study was available only in 264 infants. Missing data: 22 infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 264
Participants
  Platelet count <100.000/uL | 124
  Platelet count >100,000uL | 140

6. Secondary Outcome: Number of Subjects With INR ≥1.4.
Description: To describe the number of study subjects who experienced an INR ≥1.4 anytime during the duration of the study.
Time Frame: as for outcome 1
Population: Out of 286 infants enrolled in the study, weight at the end of study was available only in 248 infants. Missing data: 38 infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 248
Participants
  INR ≥ 1.4 | 75
  INR ≤ 1.4 | 173

7. Secondary Outcome: Number of Study Subjects Who Experienced a Blood Stream Infection
Description: To describe the number of study subjects who experienced a bloodstream infection during the duration of the study.
  Bloodstream infection as defined by detection by the culture of bacteria or fungus from the blood.
Time Frame: as for outcome 1
Population: Out of 286 infants enrolled in the study, weight at the end of study was available only in 283 infants. Missing data: 3 infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 283
Participants
  Blood stream infection | 88
  No BSI | 195

8. Secondary Outcome: Liver or Multi-visceral Transplant
Description: To describe the number and percentage of infants who required liver or multi-visceral transplant.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 286
Participants | 2

9. Secondary Outcome: All-cause Mortality up to Hospital Discharge
Description: To describe number and percentage of infants who died secondary to any cause, related or unrelated to Fish Oil Emulsion.
Time Frame: Anytime from initiation of study to discharge from the hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Emulsion Arm
Number analyzed (Participants) | 286
Participants | 40

ADVERSE EVENTS:
Time Frame: From initiation to end of study (End of Study : Discontinuation of Fish Oil Emulsion, Death, Transplant, or Discharge from the hospital, whichever is achieved first, up to 5 years).
Groups:
- Fish Oil Emulsion Arm: Once eligible, Soybean Oil Emulsion was discontinued and Fish Oil Emulsion was commenced at 1 g/kg/d. Fish Oil Emulsion was provided as an infusion over 18-24 hours a day. Fish Oil Emulsion was provided in a dedicated peripheral or central venous access.
  Any cause mortality prior to the End of Study
Arm/Group | Fish Oil Emulsion Arm
All-Cause Mortality (participants affected / at risk) | 30/286
Serious Adverse Events (participants affected / at risk) | 88/286
Other Adverse Events (participants affected / at risk) | 148/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fish Oil Emulsion Arm (N=286)
Blood Stream Infection (Infections and infestations) | 88
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fish Oil Emulsion Arm (N=286)
GGT>200 U/L (Hepatobiliary disorders) | 146
INR ≥ 1.4 (Blood and lymphatic system disorders) | 75

LIMITATIONS AND CAVEATS:
The study protocol was terminated early following the FDA approval of the Fish Oil Emulsion (Omegaven) as as source of nutrition in infants with parenteral nutrition associated cholestasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT00738101/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT00738101/ICF_001.pdf